CLINICAL TRIAL: NCT06736158
Title: Early Genomic Testing for Inherited Bleeding Disorders in Patients Without a Diagnosis After First Line Testing: a Randomized Controlled Trial
Brief Title: Early Genomic Testing for Inherited Bleeding Disorders
Acronym: GT4BD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Unity Health Toronto (Other); The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Dr. Paula James, Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4909; RDP-193724 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Bleeding Disorder
Keywords: blood coagulation disorders; bleeding disorder
MeSH Terms: conditions — Hemostatic Disorders; Blood Coagulation Disorders | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Genomic Testing Diagnostic Pathway (Experimental): Participants will receive early genomic testing in addition to standard diagnostic testing.
  Interventions: Genetic: Genetic testing for inherited bleeding disorders
- Standard Diagnostic Pathway (No Intervention): Participants will receive standard diagnostic testing with the option of receiving genomic testing after 12 months.

INTERVENTIONS:
Genetic: Genetic testing for inherited bleeding disorders — Gene panel for bleeding: This analysis will look at a list of genes known to be associated with rare coagulation, platelet, connective tissue, and bleeding disorders. There are currently 318 genes on the panel however this list may be updated throughout the study. Genes of study include those on the the International Society of Thrombosis and Haemostasis (ISTH) TIER-1 (the first group of genes are the diagnostic-grade) and TIER-2 gene list, as well as additional genes identified in published research.
  Arms: Early Genomic Testing Diagnostic Pathway

SUMMARY:
The investigators aim to test the introduction of genomic testing early in the diagnostic pathway for inherited bleeding disorders in patients who have not received a diagnosis after first-line testing.

The goal of this clinical trial is to test the introduction of genomic testing early in the diagnostic pathway for patients referred to Hematology for a suspected inherited bleeding disorder. The main questions it aims to answer are:

1. Does adding early genomic testing increase the number of patients who are diagnosed?
2. Does adding early genomic testing decrease the overall time to diagnosis?
3. Is it cost-effective to include early genomic testing in the diagnostic pathway?

The investigators will compare with a control group of participants who are receiving standard care (no early genomic testing).

Participants will randomized to a standardized diagnostic testing plus early genomic testing group or to the standardized diagnostic testing group only (with the possibility of being offered genomic testing after 1 year in the study).

DETAILED DESCRIPTION:
With the current standardized diagnostic testing process up to 50% of people referred with significant bleeding symptoms will be classified as bleeding disorder of unknown cause (BDUC), defined as those with a positive bleeding score but in whom all current diagnostic test results are repeatedly normal. Incorporating genomic testing early in the diagnostic pathway could significantly improve diagnostic yield, reduce diagnostic delay, alleviate patient anxiety, and allow for more prompt symptom recognition and targeted treatment.

ELIGIBILITY:
Inclusion Criteria:

* New patient referred for abnormal bleeding.
* Hemostasis expert clinician determined abnormal bleeding history AND family history of bleeding
* OR no family history of bleeding but hemostasis expert clinician determined severe bleeding history.

Exclusion Criteria:

* Prior diagnosis of an inherited bleeding disorder.
* Acquired cause of bleeding (i.e., medication known to cause bleeding, significant renal or hepatic disease)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | One year
  Defined as the proportion of patients who achieve a final diagnosis at one year.

SECONDARY OUTCOMES:
Time to diagnosis | One year
  The amount of time in weeks and/or months between initial Hematology visit and achieving a diagnosis of an inherited bleeding disorder
Patient Burden | One year
  This will be captured by patient reported survey. Will include data on: number of appointments for diagnosis, number of blood draws, travel (distance, mode, associated costs) and productivity loss questions (e.g. time spent away from work, wages lost, child/elder care costs).
Health Related Quality of Life | One year
  Will be determined using the PROMIS (Patient Reported Outcome Measurement Information System) Profile CAT (Computer Adaptive Testing) v1.0 - 29 for participants 18 and older, and the PROMIS Pediatric Profile GenPop (General Population) v3.0 - Profile-25 for participants 12-17. Each section consists of four items with five-point descriptive scales, except for pain intensity which has a 0-10 numerical rating scale. The sum of the item responses for each multi-item category is converted to a T-score where a score of 50 is the average for the US general population with a standard deviation of 10. Higher scores represent more of something. Therefore, for physical function, higher scores represent better health whereas for anxiety, higher scores represent poorer health.
Cost-effectiveness analysis | 2 years
  Will be measured by estimating the cost-effectiveness of the early genomic testing pathway compared with the standard diagnostic pathway (cost per diagnosis). This will be done by calculating the costs for each pathway along with the number of cases detected.
Budget Impact Analysis | 2 years
  Economic Impact will be measured by a budget impact analysis. This will be conducted from the healthcare system's perspective using standard techniques. In this model-based analysis, the incremental cost of testing for both the control and intervention arm will be determined, which will allow for detailed analysis on the economic impact of inserting genomic testing at different time points along the diagnostic algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Paula D James, MD, FRCPC, Principal Investigator — Queen's University
Locations (3):
- Canada (3):
  - Queen's University/Kingston Health Sciences Centre, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Unity Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
all (Individual Participant Data) IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be available once manuscript is accepted for publication and will be available indefinitely.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)

REFERENCES:
- [Background] Elbatarny M, Mollah S, Grabell J, Bae S, Deforest M, Tuttle A, Hopman W, Clark DS, Mauer AC, Bowman M, Riddel J, Christopherson PA, Montgomery RR; Zimmerman Program Investigators; Rand ML, Coller B, James PD. Normal range of bleeding scores for the ISTH-BAT: adult and pediatric data from the merging project. Haemophilia. 2014 Nov;20(6):831-5. doi: 10.1111/hae.12503. Epub 2014 Sep 6. PMID 25196510
- [Background] Castle D, Desborough MJR, Kemp M, Lowe G, Thomas W, Obaji S. Outcomes and management of pregnancy in women with bleeding disorder of unknown cause. J Thromb Haemost. 2022 Nov;20(11):2519-2525. doi: 10.1111/jth.15871. Epub 2022 Sep 21. PMID 36053176
- [Background] Arya S, Wilton P, Page D, Boma-Fischer L, Floros G, Winikoff R, Teitel J, Dainty K, Sholzberg M. "Everything was blood when it comes to me": Understanding the lived experiences of women with inherited bleeding disorders. J Thromb Haemost. 2020 Dec;18(12):3211-3221. doi: 10.1111/jth.15102. Epub 2020 Oct 21. PMID 32979008
- [Background] Andres O, Konig EM, Althaus K, Bakchoul T, Bugert P, Eber S, Knofler R, Kunstmann E, Manukjan G, Meyer O, Strauss G, Streif W, Thiele T, Wiegering V, Klopocki E, Schulze H; THROMKIDplus Study Group of the Society of Paediatric Oncology Haematology (Gesellschaft fur Padiatrische Onkologie und Hamatologie, GPOH) and the Society of Thrombosis Haemostasis Research (Gesellschaft fur Thrombose- und Hamostaseforschung, GTH). Use of Targeted High-Throughput Sequencing for Genetic Classification of Patients with Bleeding Diathesis and Suspected Platelet Disorder. TH Open. 2018 Dec 30;2(4):e445-e454. doi: 10.1055/s-0038-1676813. eCollection 2018 Oct. PMID 31249973
- [Background] Downes K, Borry P, Ericson K, Gomez K, Greinacher A, Lambert M, Leinoe E, Noris P, Van Geet C, Freson K; Subcommittee on Genomics in Thrombosis, Hemostasis. Clinical management, ethics and informed consent related to multi-gene panel-based high throughput sequencing testing for platelet disorders: Communication from the SSC of the ISTH. J Thromb Haemost. 2020 Oct;18(10):2751-2758. doi: 10.1111/jth.14993. PMID 33079472
- [Background] Kim SH, Kim SO, Lee SI, Jo MW. Deriving a mapping algorithm for converting SF-36 scores to EQ-5D utility score in a Korean population. Health Qual Life Outcomes. 2014 Sep 24;12:145. doi: 10.1186/s12955-014-0145-9. PMID 25248494
- [Background] Briggs A, Sculpher M, Claxton K. Decision modelling for health economic evaluation. Oup Oxford; 2006.
- [Background] Sullivan SD, Mauskopf JA, Augustovski F, Jaime Caro J, Lee KM, Minchin M, Orlewska E, Penna P, Rodriguez Barrios JM, Shau WY. Budget impact analysis-principles of good practice: report of the ISPOR 2012 Budget Impact Analysis Good Practice II Task Force. Value Health. 2014 Jan-Feb;17(1):5-14. doi: 10.1016/j.jval.2013.08.2291. Epub 2013 Dec 13. PMID 24438712
- [Background] Drummond MF, Sculpher MJ, Claxton K, Stoddart GL, Torrance GW. Methods for the economic evaluation of health care programmes. Oxford university press; 2015.
- [Background] Miller DT, Lee K, Abul-Husn NS, Amendola LM, Brothers K, Chung WK, Gollob MH, Gordon AS, Harrison SM, Hershberger RE, Klein TE, Richards CS, Stewart DR, Martin CL; ACMG Secondary Findings Working Group. Electronic address: documents@acmg.net. ACMG SF v3.1 list for reporting of secondary findings in clinical exome and genome sequencing: A policy statement of the American College of Medical Genetics and Genomics (ACMG). Genet Med. 2022 Jul;24(7):1407-1414. doi: 10.1016/j.gim.2022.04.006. Epub 2022 Jun 17. No abstract available. PMID 35802134
- [Background] Halldorsson BV, Eggertsson HP, Moore KHS, Hauswedell H, Eiriksson O, Ulfarsson MO, Palsson G, Hardarson MT, Oddsson A, Jensson BO, Kristmundsdottir S, Sigurpalsdottir BD, Stefansson OA, Beyter D, Holley G, Tragante V, Gylfason A, Olason PI, Zink F, Asgeirsdottir M, Sverrisson ST, Sigurdsson B, Gudjonsson SA, Sigurdsson GT, Halldorsson GH, Sveinbjornsson G, Norland K, Styrkarsdottir U, Magnusdottir DN, Snorradottir S, Kristinsson K, Sobech E, Jonsson H, Geirsson AJ, Olafsson I, Jonsson P, Pedersen OB, Erikstrup C, Brunak S, Ostrowski SR; DBDS Genetic Consortium; Thorleifsson G, Jonsson F, Melsted P, Jonsdottir I, Rafnar T, Holm H, Stefansson H, Saemundsdottir J, Gudbjartsson DF, Magnusson OT, Masson G, Thorsteinsdottir U, Helgason A, Jonsson H, Sulem P, Stefansson K. The sequences of 150,119 genomes in the UK Biobank. Nature. 2022 Jul;607(7920):732-740. doi: 10.1038/s41586-022-04965-x. Epub 2022 Jul 20. PMID 35859178
- [Background] Gudmundsson S, Singer-Berk M, Watts NA, Phu W, Goodrich JK, Solomonson M; Genome Aggregation Database Consortium; Rehm HL, MacArthur DG, O'Donnell-Luria A. Variant interpretation using population databases: Lessons from gnomAD. Hum Mutat. 2022 Aug;43(8):1012-1030. doi: 10.1002/humu.24309. Epub 2021 Dec 16. PMID 34859531
- [Background] Richards S, Aziz N, Bale S, Bick D, Das S, Gastier-Foster J, Grody WW, Hegde M, Lyon E, Spector E, Voelkerding K, Rehm HL; ACMG Laboratory Quality Assurance Committee. Standards and guidelines for the interpretation of sequence variants: a joint consensus recommendation of the American College of Medical Genetics and Genomics and the Association for Molecular Pathology. Genet Med. 2015 May;17(5):405-24. doi: 10.1038/gim.2015.30. Epub 2015 Mar 5. PMID 25741868
- [Background] Rydz N, Leggo J, Tinlin S, James P, Lillicrap D. The Canadian "National Program for hemophilia mutation testing" database: a ten-year review. Am J Hematol. 2013 Dec;88(12):1030-4. doi: 10.1002/ajh.23557. Epub 2013 Sep 9. PMID 23913812
- [Background] Sivapalaratnam S, Collins J, Gomez K. Diagnosis of inherited bleeding disorders in the genomic era. Br J Haematol. 2017 Nov;179(3):363-376. doi: 10.1111/bjh.14796. Epub 2017 Jun 14. PMID 28612396
- [Background] Gomez K. Advances in the diagnosis of heritable platelet disorders. Blood Rev. 2022 Nov;56:100972. doi: 10.1016/j.blre.2022.100972. Epub 2022 May 16. PMID 35595614
- [Background] Van Laer C, Jacquemin M, Baert S, Labarque V, Thys C, Vanassche T, Van Geet C, Verhamme P, Willekens K, Corveleyn A, Peerlinck K, Freson K. Clinical application of multigene panel testing for bleeding, thrombotic, and platelet disorders: a 3-year Belgian experience. J Thromb Haemost. 2023 Apr;21(4):887-895. doi: 10.1016/j.jtha.2022.12.007. Epub 2022 Dec 22. PMID 36696193
- [Background] Saes JL, Simons A, de Munnik SA, Nijziel MR, Blijlevens NMA, Jongmans MC, van der Reijden BA, Smit Y, Brons PP, van Heerde WL, Schols SEM. Whole exome sequencing in the diagnostic workup of patients with a bleeding diathesis. Haemophilia. 2019 Jan;25(1):127-135. doi: 10.1111/hae.13638. Epub 2018 Nov 15. PMID 30431218
- [Background] Andersson NG, Rossing M, Fager Ferrari M, Gabrielaite M, Leinoe E, Ljung R, Martensson A, Norstrom E, Zetterberg E. Genetic screening of children with suspected inherited bleeding disorders. Haemophilia. 2020 Mar;26(2):314-324. doi: 10.1111/hae.13948. Epub 2020 Feb 26. PMID 32100410
- [Background] Leinoe E, Zetterberg E, Kinalis S, Ostrup O, Kampmann P, Norstrom E, Andersson N, Klintman J, Qvortrup K, Nielsen FC, Rossing M. Application of whole-exome sequencing to direct the specific functional testing and diagnosis of rare inherited bleeding disorders in patients from the Oresund Region, Scandinavia. Br J Haematol. 2017 Oct;179(2):308-322. doi: 10.1111/bjh.14863. Epub 2017 Jul 27. PMID 28748566
- [Background] Stefanucci L, Collins J, Sims MC, Barrio-Hernandez I, Sun L, Burren OS, Perfetto L, Bender I, Callahan TJ, Fleming K, Guerrero JA, Hermjakob H, Martin MJ, Stephenson J, Paneerselvam K, Petrovski S, Porras P, Robinson PN, Wang Q, Watkins X, Frontini M, Laskowski RA, Beltrao P, Di Angelantonio E, Gomez K, Laffan M, Ouwehand WH, Mumford AD, Freson K, Carss K, Downes K, Gleadall N, Megy K, Bruford E, Vuckovic D. The effects of pathogenic and likely pathogenic variants for inherited hemostasis disorders in 140 214 UK Biobank participants. Blood. 2023 Dec 14;142(24):2055-2068. doi: 10.1182/blood.2023020118. PMID 37647632
- [Background] Vincent LM, Tran S, Livaja R, Bensend TA, Milewicz DM, Dahlback B. Coagulation factor V(A2440G) causes east Texas bleeding disorder via TFPIalpha. J Clin Invest. 2013 Sep;123(9):3777-87. doi: 10.1172/JCI69091. Epub 2013 Aug 27. PMID 23979162
- [Background] Langdown J, Luddington RJ, Huntington JA, Baglin TP. A hereditary bleeding disorder resulting from a premature stop codon in thrombomodulin (p.Cys537Stop). Blood. 2014 Sep 18;124(12):1951-6. doi: 10.1182/blood-2014-02-557538. Epub 2014 Jul 21. PMID 25049278
- [Background] Mehic D, Tolios A, Hofer S, Ay C, Haslacher H, Rejto J, Ouwehand WH, Downes K, Haimel M, Pabinger I, Gebhart J. Elevated levels of tissue factor pathway inhibitor in patients with mild to moderate bleeding tendency. Blood Adv. 2021 Jan 26;5(2):391-398. doi: 10.1182/bloodadvances.2020003464. PMID 33496735
- [Background] Mehic D, Tolios A, Hofer S, Ay C, Haslacher H, Downes K, Haimel M, Pabinger I, Gebhart J. Thrombomodulin in patients with mild to moderate bleeding tendency. Haemophilia. 2021 Nov;27(6):1028-1036. doi: 10.1111/hae.14433. Epub 2021 Oct 10. PMID 34628704
- [Background] Thomas W, Downes K, Desborough MJR. Bleeding of unknown cause and unclassified bleeding disorders; diagnosis, pathophysiology and management. Haemophilia. 2020 Nov;26(6):946-957. doi: 10.1111/hae.14174. Epub 2020 Oct 23. PMID 33094877
- [Background] Thomas W. The natural history of bleeding disorder of unknown cause. J Thromb Haemost. 2023 Jul;21(7):1747-1749. doi: 10.1016/j.jtha.2023.03.025. No abstract available. PMID 37330263
- [Background] Gebhart J, Hofer S, Panzer S, Quehenberger P, Sunder-Plassmann R, Hoermann G, Eigenbauer E, Haslacher H, Kepa S, Kyrle PA, Eichinger S, Knobl P, Eischer L, Mannhalter C, Ay C, Pabinger I. High proportion of patients with bleeding of unknown cause in persons with a mild-to-moderate bleeding tendency: Results from the Vienna Bleeding Biobank (VIBB). Haemophilia. 2018 May;24(3):405-413. doi: 10.1111/hae.13422. Epub 2018 Feb 1. PMID 29388750
- [Background] Toole JJ, Knopf JL, Wozney JM, Sultzman LA, Buecker JL, Pittman DD, Kaufman RJ, Brown E, Shoemaker C, Orr EC, et al. Molecular cloning of a cDNA encoding human antihaemophilic factor. Nature. 1984 Nov 22-28;312(5992):342-7. doi: 10.1038/312342a0. PMID 6438528
- [Background] Kurachi K, Davie EW. Isolation and characterization of a cDNA coding for human factor IX. Proc Natl Acad Sci U S A. 1982 Nov;79(21):6461-4. doi: 10.1073/pnas.79.21.6461. PMID 6959130
- [Background] Choo KH, Gould KG, Rees DJ, Brownlee GG. Molecular cloning of the gene for human anti-haemophilic factor IX. Nature. 1982 Sep 9;299(5879):178-80. doi: 10.1038/299178a0. PMID 6287289
- [Background] MacDonald S, Wright A, Beuche F, Downes K, Besser M, Symington E, Kelly A, Thomas W. Characterization of a large cohort of patients with unclassified bleeding disorder; clinical features, management of haemostatic challenges and use of global haemostatic assessment with proposed recommendations for diagnosis and treatment. Int J Lab Hematol. 2020 Apr;42(2):116-125. doi: 10.1111/ijlh.13124. Epub 2019 Nov 20. PMID 31747136
- [Background] Mehic D, Schwarz S, Shulym I, Ay C, Pabinger I, Gebhart J. Health-related quality of life is impaired in bleeding disorders of unknown cause: results from the Vienna Bleeding Biobank. Res Pract Thromb Haemost. 2023 Aug 22;7(6):102176. doi: 10.1016/j.rpth.2023.102176. eCollection 2023 Aug. PMID 37720482
- [Background] Gilbert L, Paroskie A, Gailani D, Debaun MR, Sidonio RF. Haemophilia A carriers experience reduced health-related quality of life. Haemophilia. 2015 Nov;21(6):761-5. doi: 10.1111/hae.12690. Epub 2015 Apr 30. PMID 25930174
- [Background] Chaigneau M, James PD. Approach to the Patient with Bleeding. Hematol Oncol Clin North Am. 2021 Dec;35(6):1039-1049. doi: 10.1016/j.hoc.2021.07.001. Epub 2021 Sep 15. PMID 34535288
- [Background] Federici AB, Bucciarelli P, Castaman G, Mazzucconi MG, Morfini M, Rocino A, Schiavoni M, Peyvandi F, Rodeghiero F, Mannucci PM. The bleeding score predicts clinical outcomes and replacement therapy in adults with von Willebrand disease. Blood. 2014 Jun 26;123(26):4037-44. doi: 10.1182/blood-2014-02-557264. Epub 2014 Apr 30. PMID 24786773
- [Background] Casey LJ, Tuttle A, Grabell J, Hopman W, Moorehead PC, Blanchette VS, Wu JK, Steele M, Klaassen RJ, Silva M, Rand ML, James PD. Generation and optimization of the self-administered pediatric bleeding questionnaire and its validation as a screening tool for von Willebrand disease. Pediatr Blood Cancer. 2017 Oct;64(10). doi: 10.1002/pbc.26588. Epub 2017 Apr 28. PMID 28453185
- [Background] Deforest M, Grabell J, Albert S, Young J, Tuttle A, Hopman WM, James PD. Generation and optimization of the self-administered bleeding assessment tool and its validation as a screening test for von Willebrand disease. Haemophilia. 2015 Sep;21(5):e384-8. doi: 10.1111/hae.12747. Epub 2015 Jul 14. PMID 26179127
- [Background] Rodeghiero F, Tosetto A, Abshire T, Arnold DM, Coller B, James P, Neunert C, Lillicrap D; ISTH/SSC joint VWF and Perinatal/Pediatric Hemostasis Subcommittees Working Group. ISTH/SSC bleeding assessment tool: a standardized questionnaire and a proposal for a new bleeding score for inherited bleeding disorders. J Thromb Haemost. 2010 Sep;8(9):2063-5. doi: 10.1111/j.1538-7836.2010.03975.x. No abstract available. PMID 20626619
- [Background] Srivastava A, Santagostino E, Dougall A, Kitchen S, Sutherland M, Pipe SW, Carcao M, Mahlangu J, Ragni MV, Windyga J, Llinas A, Goddard NJ, Mohan R, Poonnoose PM, Feldman BM, Lewis SZ, van den Berg HM, Pierce GF; WFH Guidelines for the Management of Hemophilia panelists and co-authors. WFH Guidelines for the Management of Hemophilia, 3rd edition. Haemophilia. 2020 Aug;26 Suppl 6:1-158. doi: 10.1111/hae.14046. Epub 2020 Aug 3. No abstract available. PMID 32744769
- [Background] James PD, Connell NT, Ameer B, Di Paola J, Eikenboom J, Giraud N, Haberichter S, Jacobs-Pratt V, Konkle B, McLintock C, McRae S, R Montgomery R, O'Donnell JS, Scappe N, Sidonio R, Flood VH, Husainat N, Kalot MA, Mustafa RA. ASH ISTH NHF WFH 2021 guidelines on the diagnosis of von Willebrand disease. Blood Adv. 2021 Jan 12;5(1):280-300. doi: 10.1182/bloodadvances.2020003265. PMID 33570651
- [Background] Bolton-Maggs PH, Chalmers EA, Collins PW, Harrison P, Kitchen S, Liesner RJ, Minford A, Mumford AD, Parapia LA, Perry DJ, Watson SP, Wilde JT, Williams MD; UKHCDO. A review of inherited platelet disorders with guidelines for their management on behalf of the UKHCDO. Br J Haematol. 2006 Dec;135(5):603-33. doi: 10.1111/j.1365-2141.2006.06343.x. PMID 17107346
- [Background] Atiq F, Saes JL, Punt MC, van Galen KPM, Schutgens REG, Meijer K, Cnossen MH, Laros-Van Gorkom BAP, Peters M, Nieuwenhuizen L, Kruip MJHA, de Meris J, van der Bom JG, van der Meer FJM, Fijnvandraat K, Kruis IC, van Heerde WL, Eikenboom HCJ, Leebeek FWG, Schols SEM; WiN, RBiN and TiN study groups. Major differences in clinical presentation, diagnosis and management of men and women with autosomal inherited bleeding disorders. EClinicalMedicine. 2021 Jan 29;32:100726. doi: 10.1016/j.eclinm.2021.100726. eCollection 2021 Feb. PMID 33554093
- [Background] Pruthi RK. Testing strategies used in the diagnosis of rare inherited bleeding disorders. Expert Rev Hematol. 2023 Jun;16(6):451-465. doi: 10.1080/17474086.2023.2211257. Epub 2023 May 8. PMID 37144355
- [Background] Richter T, Nestler-Parr S, Babela R, Khan ZM, Tesoro T, Molsen E, Hughes DA; International Society for Pharmacoeconomics and Outcomes Research Rare Disease Special Interest Group. Rare Disease Terminology and Definitions-A Systematic Global Review: Report of the ISPOR Rare Disease Special Interest Group. Value Health. 2015 Sep;18(6):906-14. doi: 10.1016/j.jval.2015.05.008. Epub 2015 Aug 18. PMID 26409619
- [Background] Quiroga T, Goycoolea M, Panes O, Aranda E, Martinez C, Belmont S, Munoz B, Zuniga P, Pereira J, Mezzano D. High prevalence of bleeders of unknown cause among patients with inherited mucocutaneous bleeding. A prospective study of 280 patients and 299 controls. Haematologica. 2007 Mar;92(3):357-65. doi: 10.3324/haematol.10816. PMID 17339185
- [Background] Srivastava A. Diagnosis of haemophilia and other inherited bleeding disorders - Is a new paradigm needed? Haemophilia. 2021 Feb;27 Suppl 3:14-20. doi: 10.1111/hae.14042. Epub 2020 Jun 14. PMID 32537805
- [Background] Chaigneau M, Bowman M, Grabell J, Conboy M, Johnson A, Thorpe K, Guerin A, Dinchong R, Paterson A, Good D, Mahar A, Callum J, Wheaton L, Leung J, Khalife R, Sholzberg M, Lillicrap D, James PD. Genomic testing for bleeding disorders (GT4BD): protocol for a randomised controlled trial evaluating the introduction of whole genome sequencing early in the diagnostic pathway for patients with inherited bleeding disorders as compared with standard of care. BMJ Open. 2025 Apr 17;15(4):e102041. doi: 10.1136/bmjopen-2025-102041. PMID 40246558